CLINICAL TRIAL: NCT01868750
Title: A Phase 2, Placebo-controlled, Randomized Study to Evaluate the Effect of Pre-operative Vitamin D Supplementation on Hypocalcemia Following Total or Near-total Thyroidectomy
Brief Title: Phase II Pre-operative Vitamin D Supplementation to Prevent Post-thyroidectomy Hypocalcemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: David Shonka, MD (Other)
Responsible Party: Sponsor-Investigator, David Shonka, MD, Assistant Professor, University of Virginia
Organization: University of Virginia (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 16544
Record Dates: First submitted 2013-05-30; First posted 2013-06-04 (Estimated); Last update posted 2021-10-12 (Actual); Status verified 2021-10

CONDITIONS: Thyroid Nodules; Hypocalcemia
MeSH Terms: conditions — Thyroid Nodule; Hypocalcemia | interventions — Calcitriol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Vitamin D (Calcitriol) (Active Comparator): Calcitriol, 1.0ug twice daily for 7 days prior to surgery
  Interventions: Dietary Supplement: Calcitriol
- Control (Placebo Comparator): Placebo pill taken twice daily for 7 days prior to surgery
  Interventions: Dietary Supplement: Control Pill

INTERVENTIONS:
Dietary Supplement: Calcitriol — 1.0ug twice daily for 7 days before surgery
  Arms: Vitamin D (Calcitriol)
Dietary Supplement: Control Pill — placebo pill taken twice daily for 7 days before surgery
  Arms: Control

SUMMARY:
One of the major side effects of surgery to remove the thyroid gland is transient (lasting for a short time) low calcium levels in the blood, or "hypocalcemia." Low calcium levels can cause symptoms such as numbness around the mouth, tingling or cramping in the hands and feet, severe muscle spasms, inability to breathe, or heart rhythm (heart beat) abnormalities. Severe symptoms are life threatening, so it is important to start the management of these symptoms in the hospital. Treating low calcium levels sometimes require patients to spend a few extra days in the hospital.

The human body needs vitamin D to function and stay healthy. Vitamin D helps the body get the calcium needed to make strong bones and teeth. The purpose of this study is to determine if taking vitamin D before surgery to remove the thyroid gland affects whether or not you may have low calcium levels after your surgery and to test the hypothesis that those who are given the Vitamin D before surgery will have decreased hypocalcemia and a shortened hospital stay.

ELIGIBILITY:
Inclusion Criteria:

* Patient referred for thyroidectomy
* Agreement to use contraception prior to and during the study

Exclusion Criteria:

* Hypercalcemia (>10.5mg/dL)
* Chronic kidney or parathyroid disease
* Cardiac or Central Nervous System disease
* Pregnant or breastfeeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Estimated)
Dates: Start 2013-05; Primary Completion 2021-07-08 (Actual); Study Completion 2021-07-08 (Actual)

PRIMARY OUTCOMES:
Measure of Serum Calcium Levels | 2-5 days after surgery
  Serum calcium levels will be evaluated at routine intervals to identify incidences of hypocalcemia

SECONDARY OUTCOMES:
Evidence of Hypocalcemia | 2-5 days after surgery
  Measuring hypocalcemia symptoms, requirements for IV calcium, and extended hospital stay

CONTACTS AND LOCATIONS:
Overall Officials: David C Shonka, MD, Principal Investigator — University of Virginia
Locations (1):
- University of Virginia, Charlottesville, Virginia, United States